CLINICAL TRIAL: NCT03289416
Title: Efficacy of Bone Marrow Aspirate Concentrate Compared With Platelet Rich Plasma for the Treatment of Symptomatic Knee Osteoarthritis: A Randomized, Controlled Clinical Trial
Brief Title: Bone Marrow Aspirate Compared to Platelet Rich Plasma for Treating Knee Osteoarthritis
Acronym: EmCyte
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrews Research & Education Foundation (Other)
Collaborators: EmCyte Corporation (Industry); BioSciences Research Associates, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EmCyte
Record Dates: First submitted 2017-09-18; First posted 2017-09-21 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee; osteoarthritis; platelet rich plasma (PRP); bone marrow concentrate (BMC)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either a PRP intervention group or the BMC intervention group. Knee pain and function outcomes of enrolled patients in the two groups will be compared to determine which treatment is more effective in treating knee osteoarthritis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma (PRP) (Other): Blood will be drawn from the patient using the Pure PRP II system into a syringe with anticoagulant (sodium citrate). 1 mL of blood will be separated and sent to a lab for analysis. Remaining blood will be separated into a single concentrating device and centrifuged to separate red blood cells from plasma and platelets. The plasma and platelets will be separated off with a syringe and re-centrifuged to separate the platelets from the plasma. 1 mL will be separated and sent to a lab for analysis leaving 6 mL for injection. Both the 1 mL of blood and the 1 mL of PRP will be sent to an independent lab to undergo analysis for CBC, TNC, human CD34+ hematopoietic stem/progenitor cell assay and CFU-F. Physician will then inject the PRP into the affected knee joint.
  Interventions: Combination Product: Pure PRP II
- Bone Marrow Concentrate (BMC) (Other): Bone marrow will be harvested from the posterior iliac crest using the PureBMC system. 50 mL of bone marrow will be drawn into one syringe containing 10 mL of sodium citrate. Marrow will be filtered and centrifuged for separation of the bone marrow concentrate. Plasma and cell concentrate will be separated off with two syringes and re-centrifuged to separate the cell concentrate from the plasma. After plasma is drawn off, BMC will be drawn into a syringe for injection into affected knee. BMC production procedure results in 7 mL of product and 1 mL will be separated and sent to a lab for analysis. Both 1 mL of BMA and 1 mL of BMC will be sent to an independent lab to undergo analysis for CBC, TNC, human CD34+ hematopoietic stem/progenitor cell assay and CFU-F.
  Interventions: Combination Product: PureBMC

INTERVENTIONS:
Combination Product: Pure PRP II — The Pure PRP II system will be used to collect and concentrate blood into platelet rich plasma that will be injected into the knee.
  Other Names: GS60-PURE-II
  Arms: Platelet Rich Plasma (PRP)
Combination Product: PureBMC — The PureBMC system will be used to collect and concentrate bone marrow aspirate into bone marrow concentrate that will be injected into the knee.
  Other Names: BC60-PURE
  Arms: Bone Marrow Concentrate (BMC)

SUMMARY:
This study is intended to compare whether bone marrow aspirate concentrate or platelet rich plasma injections is more effective in treating knee osteoarthritis.

DETAILED DESCRIPTION:
While PRP shows promise in helping restore function to these patients, there are still concerns with PRP's long term outcomes. Another option that has become more popular for physicians treating this debilitation condition is bone marrow aspirate concentrate (BMA), which use's undifferentiated cells found in the bone marrow to promote healing and tissue regeneration. These cells have the ability to replicate into a multiple different tissue types. With BMA, the marrow is concentrated provide better healing of the damaged tissue and aid in growth and repair. The full benefits of BMA are still unknown, but studies have shown the treatment can reduce swelling, relieve pain, and improve healing in articular cartilage and bone grafts.

Autologous BMA has shown promising clinical potential as a therapeutic agent in regenerative medicine, including the treatment of osteoarthritis and cartilage defects, and the clinical efficacy platelet rich plasma has been documented to alleviate symptoms related to knee osteoarthritis. However, randomized, prospective comparison of the two techniques has not been reported in the literature and long term follow-up for both treatments is limited, and especially limited in the use of BMA for osteoarthritis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-80 years
* Knee osteoarthritis
* Subjects must present with pain or swelling to target knee for at least 4 months
* Kellgren-Lawrence score between 1 and 3 upon x-ray evaluation
* Must be willing and able to provide informed consent
* Willing and able to return for scheduled follow-up visits

Exclusion Criteria:

* Major mechanical axis deviation of more than 50% into either compartment (varus or valgus )
* Have had a corticosteroid injection within 3 months or a hyaluronic acid injection within 6 months
* History of the following medical conditions:
* diabetes
* autoimmune disorders
* disorders requiring immunosuppression
* rheumatoid arthritis
* hemophilic arthropathy
* infectious arthritis
* Charcot's knee
* Paget's disease of the femur or tibia
* Cancer
* Ongoing infectious disease
* Significant cardiovascular, renal or hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Hackel, MD, Principal Investigator — Andrews Institute for Orthopaedic & Sports Medicine
Locations (1):
- Andrews Research & Education Foundation, Gulf Breeze, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hootman JM, Helmick CG. Projections of US prevalence of arthritis and associated activity limitations. Arthritis Rheum. 2006 Jan;54(1):226-9. doi: 10.1002/art.21562. PMID 16385518
- [Background] Spakova T, Rosocha J, Lacko M, Harvanova D, Gharaibeh A. Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2012 May;91(5):411-7. doi: 10.1097/PHM.0b013e3182aab72. PMID 22513879
- [Background] Kon E, Mandelbaum B, Buda R, Filardo G, Delcogliano M, Timoncini A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular injection versus hyaluronic acid viscosupplementation as treatments for cartilage pathology: from early degeneration to osteoarthritis. Arthroscopy. 2011 Nov;27(11):1490-501. doi: 10.1016/j.arthro.2011.05.011. Epub 2011 Aug 10. PMID 21831567
- [Background] Cerza F, Carni S, Carcangiu A, Di Vavo I, Schiavilla V, Pecora A, De Biasi G, Ciuffreda M. Comparison between hyaluronic acid and platelet-rich plasma, intra-articular infiltration in the treatment of gonarthrosis. Am J Sports Med. 2012 Dec;40(12):2822-7. doi: 10.1177/0363546512461902. Epub 2012 Oct 25. PMID 23104611
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Li M, Zhang C, Ai Z, Yuan T, Feng Y, Jia W. [Therapeutic effectiveness of intra-knee-articular injection of platelet-rich plasma on knee articular cartilage degeneration]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2011 Oct;25(10):1192-6. Chinese. PMID 22069972
- [Background] Filardo G, Kon E, Di Martino A, Di Matteo B, Merli ML, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma vs hyaluronic acid to treat knee degenerative pathology: study design and preliminary results of a randomized controlled trial. BMC Musculoskelet Disord. 2012 Nov 23;13:229. doi: 10.1186/1471-2474-13-229. PMID 23176112
- [Background] Vaquerizo V, Plasencia MA, Arribas I, Seijas R, Padilla S, Orive G, Anitua E. Comparison of intra-articular injections of plasma rich in growth factors (PRGF-Endoret) versus Durolane hyaluronic acid in the treatment of patients with symptomatic osteoarthritis: a randomized controlled trial. Arthroscopy. 2013 Oct;29(10):1635-43. doi: 10.1016/j.arthro.2013.07.264. PMID 24075613
- [Background] Convery PN, Milligan KR, Quinn P, Scott K, Clarke RC. Low-dose intra-articular ketorolac for pain relief following arthroscopy of the knee joint. Anaesthesia. 1998 Nov;53(11):1125-9. doi: 10.1046/j.1365-2044.1998.00582.x. PMID 10023285
- [Background] Ng HP, Nordstrom U, Axelsson K, Perniola AD, Gustav E, Ryttberg L, Gupta A. Efficacy of intra-articular bupivacaine, ropivacaine, or a combination of ropivacaine, morphine, and ketorolac on postoperative pain relief after ambulatory arthroscopic knee surgery: a randomized double-blind study. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):26-33. doi: 10.1016/j.rapm.2005.09.009. PMID 16418021
- [Background] Gupta A, Axelsson K, Allvin R, Liszka-Hackzell J, Rawal N, Althoff B, Augustini BG. Postoperative pain following knee arthroscopy: the effects of intra-articular ketorolac and/or morphine. Reg Anesth Pain Med. 1999 May-Jun;24(3):225-30. doi: 10.1016/s1098-7339(99)90132-3. PMID 10338172
- [Background] Beitzel K, McCarthy MB, Cote MP, Apostolakos J, Russell RP, Bradley J, ElAttrache NS, Romeo AA, Arciero RA, Mazzocca AD. The effect of ketorolac tromethamine, methylprednisolone, and platelet-rich plasma on human chondrocyte and tenocyte viability. Arthroscopy. 2013 Jul;29(7):1164-74. doi: 10.1016/j.arthro.2013.04.006. PMID 23809450
- [Background] Hauser RA, Orlofsky A. Regenerative injection therapy with whole bone marrow aspirate for degenerative joint disease: a case series. Clin Med Insights Arthritis Musculoskelet Disord. 2013 Sep 4;6:65-72. doi: 10.4137/CMAMD.S10951. eCollection 2013. PMID 24046512
- [Background] Saw KY, Hussin P, Loke SC, Azam M, Chen HC, Tay YG, Low S, Wallin KL, Ragavanaidu K. Articular cartilage regeneration with autologous marrow aspirate and hyaluronic Acid: an experimental study in a goat model. Arthroscopy. 2009 Dec;25(12):1391-400. doi: 10.1016/j.arthro.2009.07.011. Epub 2009 Sep 17. PMID 19962065
- [Derived] Anz AW, Plummer HA, Cohen A, Everts PA, Andrews JR, Hackel JG. Bone Marrow Aspirate Concentrate Is Equivalent to Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis at 2 Years: A Prospective Randomized Trial. Am J Sports Med. 2022 Mar;50(3):618-629. doi: 10.1177/03635465211072554. PMID 35289231
- [Derived] Anz AW, Hubbard R, Rendos NK, Everts PA, Andrews JR, Hackel JG. Bone Marrow Aspirate Concentrate Is Equivalent to Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis at 1 Year: A Prospective, Randomized Trial. Orthop J Sports Med. 2020 Feb 18;8(2):2325967119900958. doi: 10.1177/2325967119900958. eCollection 2020 Feb. PMID 32118081

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Platelet Rich Plasma (PRP) | Bone Marrow Concentrate (BMC)
Started | 41 | 49
Completed | 41 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet Rich Plasma (PRP) | Bone Marrow Concentrate (BMC) | Total
Number analyzed (Participants) | 41 | 49 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (12.4) | 55.8 (11.3) | 54.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 23 | 28 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 41 | 49 | 90

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Measurements
Description: Pain score measurements utilizing patient surveys; scale 0-20 with 20 being most pain and 0 being least pain
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, and 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) | Bone Marrow Concentrate (BMC)
Number analyzed (Participants) | 41 | 49
score on a scale
  Baseline | 32.1 [26.4 to 37.9] | 35.3 [29.9 to 40.6]
  1 month | 19.5 [14.6 to 24.4] | 19.8 [15.2 to 24.3]
  3 Months | 18.2 [13.7 to 22.8] | 15.2 [11 to 19.4]
  6 Months | 16.2 [11 to 21.5] | 19.4 [14.5 to 24.3]
  9 Months | 18.4 [13.1 to 23.7] | 17.6 [12.7 to 22.6]
  12 Months | 16.8 [11.5 to 22.1] | 19.4 [14.5 to 24.3]

2. Secondary Outcome: Subjective International Knee Documentation Committee Subjective Score (IKDC)
Description: Pain score measurement utilizing patient surveys; scale is 0-100 with 0 being lowest level of function and 100 being the highest
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, and 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Platelet Rich Plasma (PRP) | Bone Marrow Concentrate (BMC)
Number analyzed (Participants) | 41 | 49
score on a scale
  Baseline | 47.4 [42.5 to 52.3] | .909 [-6.3 to 7.0]
  1 Month | 58.4 [52.5 to 64.4] | 58.5 [53 to 64.1]
  3 Months | 61.6 [56.2 to 67.1] | 63.6 [58.6 to 68.7]
  6 Months | 65 [58.5 to 71.5] | 63.7 [57.6 to 69.7]
  9 Months | 63.1 [56.3 to 69.9] | 63.7 [57.4 to 70]
  12 Months | 63.7 [57.2 to 70.1] | 64.3 [58.3 to 70.3]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Platelet Rich Plasma (PRP) | Bone Marrow Concentrate (BMC)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/41 | 2/49
Other Adverse Events (participants affected / at risk) | 0/41 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet Rich Plasma (PRP) (N=41) | Bone Marrow Concentrate (BMC) (N=49)
Patient Hospitalized due to Unrelated Ailments (General disorders) | 0 (0) | 1 (1) — Subject fell off of her horse on 3 Feb 2017 and sustained a right proximal humerus fracture. Subject was admitted to the ER at Baptist hospital in Pensacola on 3 Feb 2017, had surgery performed on 4 Feb 2017, and was discharged on 5 February 2017.
Patient Withdrawn due to Unrelated Ailments (Immune system disorders) | 0 (0) | 1 (1) — Subject called the CRC. Subject stated that they saw a doctor due to pain in their arm and it was found out that the arm was broken possibly due to multiple myeloma. Subject verbally stated over the phone desire to withdraw from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03289416/Prot_SAP_000.pdf